CLINICAL TRIAL: NCT06439355
Title: Single-center Study of Gustation in Idiopathic Parkinson's Disease and Lewy Body Disease Using Gustatory Evoked Potential Analysis
Acronym: PI-PEG
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Universitaire Dijon (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: SCHNEIDER J'InvEST-I 2023
Record Dates: First submitted 2024-05-28; First posted 2024-06-03 (Actual); Last update posted 2024-06-07 (Actual); Status verified 2024-06

CONDITIONS: Idiopathic Parkinson's Disease and Lewy Body Disease
MeSH Terms: conditions — Parkinson Disease; Lewy Body Disease | interventions — Mental Status and Dementia Tests; Nutrition Assessment

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Healthy volunteers (Active Comparator)
  Interventions: Biological: Fasting blood test; Other: Subject interview; Other: Motor assessment; Other: Neurocognitive assessment; Other: Nutritional assessment; Other: Taste tests
- Patients with Idiopathic Parkinson's Disease (IPD) of course ≤ 3 years (Experimental)
  Interventions: Biological: Fasting blood test; Other: Subject interview; Other: Motor assessment; Other: Neurocognitive assessment; Other: Nutritional assessment; Other: Taste tests
- Patients with Lewy body disease (LBD) progressing ≤ 3 years (Experimental)
  Interventions: Biological: Fasting blood test; Other: Subject interview; Other: Motor assessment; Other: Neurocognitive assessment; Other: Nutritional assessment; Other: Taste tests

INTERVENTIONS:
Biological: Fasting blood test — metabolic assays determination of food intake hormones oxidative stress and neurodegeneration marker assays
Other: Subject interview — socio-demographic data, medical and family history, treatment taken
Other: Motor assessment — MDS-UPDRS scale PART III
Other: Neurocognitive assessment — MoCA and MMSE scales
Other: Nutritional assessment — anthropometric data (weight, height, BMI, waist circumference, hip circumference, android/gynoid ratio, triceps skin fold, brachial circumference), bioelectrical impedancemetry (fat mass, lean mass, water mass and bone mass)
Other: Taste tests — Recording of PEGs in response to a sucrose solution and a free fatty acid solution (prepared beforehand)

SUMMARY:
The aim of the PI-PEG study is to explore the taste functions of the following 3 groups of participants:

* healthy volunteers
* patients with early Parkinson's disease
* patients with incipient Lewy body disease.

To this end, the results obtained from taste evoked potentials in each of the 3 groups of participants will be compared with each other and with different nutritional, motor and cognitive data.

This study could reveal a difference in cortical processing of gustatory sensory information between patients who have had idiopathic Parkinson's disease progressing for 3 years or less, and patients who have had Lewy body disease progressing for 3 years or less. Indeed, a modification of taste evoked potentials (in terms of latencies) proportional to the degree of cerebral degeneration could be observed.

ELIGIBILITY:
Inclusion Criteria:

Healthy volunteers:

* Person who has given written consent
* Adult
* Enrolled in the national register of healthy volunteers
* Fasting > 2 hours before PEG measurement
* Body Mass Index (BMI) < 30 kg/m².
* No cognitive complaints and normal neurological assessment

Patients with idiopathic Parkinson's disease:

* Person who has given written consent
* Adult
* Fasting > 2 hours before PEG measurement
* Body Mass Index (BMI) < 30 kg/m².
* Diagnostic criteria for established or probable IPD

Patients with Lewy body disease:

* Person who has given written consent
* Adult
* Fasting > 2 hours prior to PEG measurement
* Body Mass Index (BMI) < 30 kg/m².
* Diagnostic criteria for probable or possible LBD

Exclusion Criteria:

* Non-affiliated to national health insurance
* Person under legal protection (curatorship, guardianship)
* Person subject to a court order
* Pregnant, parturient or breast-feeding women
* Major unable to give consent
* MMSE score < 15 and/or MoCA < 10
* Known infection with COVID-19 in the 6 months prior to inclusion
* Active smoker (> 4 cigarettes per day on a regular basis)
* Subject with pacemaker (contraindication for bioelectrical impedancemetry)
* Diabetic (type 1 or type 2)
* Taking medication (in progress at the time of the study) that interferes with gustation

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 66 (Estimated)
Dates: Start 2024-05-27 (Actual); Primary Completion 2026-05 (Estimated); Study Completion 2026-05 (Estimated)

PRIMARY OUTCOMES:
Average latency of taste-evoked potentials | After a 2-hour fasting period

CONTACTS AND LOCATIONS:
Locations (1):
- Chu Dijon Bourgogne, Dijon, France